CLINICAL TRIAL: NCT06963879
Title: Validation Study of a New Digital Diagnostic and Treatment Test Based on Interactive Video Games for Alzheimer's Disease
Acronym: EyeAD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Braingaze (Industry)
Responsible Party: Principal Investigator, Hans Supèr, Principal Investigator, Braingaze
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID2022-139968OB-I00
Record Dates: First submitted 2025-04-22; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; MCI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BGaze Therapy MCI (Experimental): 30 Patients with Mild Cognitive Impairment for validation and 15 for therapy
  Interventions: Device: Bgaze Therapy; Diagnostic Test: Bgaze Attention Task
- BGaze Therapy AD (Experimental): 30 Patients with Early Alzheimer's Disease for validation and 15 for therapy
  Interventions: Device: Bgaze Therapy; Diagnostic Test: Bgaze Attention Task

INTERVENTIONS:
Device: Bgaze Therapy — BGaze Therapy is a digital intervention by Braingaze designed to enhance attention and memory in individuals with Alzheimer's Disease (AD) and Mild Cognitive Impairment (MCI). It uses an interactive video game controlled through eye-tracking, allowing users to play using only their gaze. The therapy is based on research linking eye vergence and pupil responses to cognitive processing-physiological markers that may indicate neurodegeneration. During gameplay, these responses are modulated, potentially inducing gamma brain oscillations associated with reduced AD pathology. Patients play at care-center for 5-10 minutes daily over two months. Equipment is provided, and both in-person and remote support ensure usability. The game adapts difficulty in real time and provides feedback to keep users engaged and stimulate cognitive function.
Diagnostic Test: Bgaze Attention Task — For the validation of diagnosis of AD with vergence method the Attention Test (B-Gaze) will be used. This is an odd ball paradigm where visual target has to be detected among blue distractors. The test consist of 100 trials of 1 second and last about 3 minutes. The task uses remote eye infra-red tracking to measure eye vergence. Subjects merely have to fixate at the computer screen during the task.

SUMMARY:
This study aims to validate a novel, non-invasive diagnostic and digital therapeutic approach for Alzheimer's Disease (AD), centered on an interactive video game called BGaze Therapy. This platform leverages eye-tracking technology to assess and potentially enhance cognitive functions, particularly attention and memory.

The diagnostic component of the study investigates the use of eye vergence responses-elicited during a visual attention task-as potential biomarkers for early AD. Specifically, the study will re-validate eye vergence by comparing response patterns among three groups: cognitively healthy older adults, individuals with Mild Cognitive Impairment (MCI), and patients with confirmed AD, based on blood biomarkers (ßA40, ßA42, pTau181, and pTau217). The diagnostic task follows an oddball paradigm, where participants must detect target images (grapes) among distractors (other fruits) across 100 one-second trials, lasting approximately three minutes. Eye vergence is recorded using remote infrared eye-tracking, while participants simply fixate on a computer screen.

The therapeutic aspect evaluates the impact of BGaze Therapy, which employs "serious games" designed to train attentional control through eye movements. The game dynamically adjusts its difficulty in real time and provides continuous feedback to enhance user engagement and learning efficacy.

Participants will undergo pre-testing-including blood biomarker analysis and standardized cognitive assessments (MMSE and MoCA)-followed by a two-month training phase at care centers using the BGaze Therapy system. Post-intervention testing will mirror the pre-test protocol to assess cognitive and neurological changes.

A total of 60 participants (30 with MCI and 30 with AD) will be recruited for the validation phase. A subsample (15 MCI and 15 AD participants) will be selected for the treatment phase.

Ultimately, this study aims to establish BGaze as a cost-effective, scalable, and non-invasive tool for the early diagnosis and treatment of Alzheimer's Disease by addressing the attentional and cognitive deficits associated with the condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older.
* Clinical diagnosis of early-stage AD or MCI based the criteria of National Institute on Aging-Alzheimer's Association.
* Capable of providing informed consent.

Exclusion Criteria:

* Severe cognitive impairment (MMSE < 10).
* Neurological conditions affecting cognition (e.g., stroke).
* Severe psychiatric disorders.
* Structural brain abnormalities (e.g., tumors) with cognitive impact.
* Significant visual impairments.
* Inability to understand or communicate in Spanish.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Beta biomarkers | Immediately after the intervention
  Measure changes in plasma ßA40 and ßA42 in pg/mL
PTau Biomarkers | Immediately after the intervention
  Measure changes in plasma PTau181 and pTau217 in pg/mL
Pupil Response | Immediately after the intervention
  Pupillary diameter in millimeters (mm) will be calculated from data obtained using eye-tracking devices.
Ocular vergence | Immediately after the intervention
  Ocular vergence in degrees (°) will be calculated from data obtained using eye-tracking devices.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) Score | Immediately after the intervention
  Score in the Montreal Cognitive Assessment (MoCA); units on a scale (0-30), with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Braingaze, Mataró, Barcelona, Spain

REFERENCES:
- [Background] Romeo A, Leonovych O, Sole Puig M, Super H. Cognitive Vergence Recorded with a Webcam-Based Eye-Tracker during an Oddball Task in an Elderly Population. Sensors (Basel). 2024 Jan 30;24(3):888. doi: 10.3390/s24030888. PMID 38339605
- [Background] Jimenez EC, Sierra-Marcos A, Romeo A, Hashemi A, Leonovych O, Bustos Valenzuela P, Sole Puig M, Super H. Altered Vergence Eye Movements and Pupil Response of Patients with Alzheimer's Disease and Mild Cognitive Impairment During an Oddball Task. J Alzheimers Dis. 2021;82(1):421-433. doi: 10.3233/JAD-201301. PMID 34024820
- [Background] Hashemi A, Leonovych O, Jiménez EC, Sierra-Marcos A, Romeo A, Valenzuala PB, et al. Classification of MCI patients using vergence eye movements and pupil responses obtained during a visual oddball test. Aging Health Res. 2023 Mar 1;3(1):100121.